CLINICAL TRIAL: NCT05697653
Title: Effect of Skin to Skin Contact on Sucking Efficiency of Newborns and Breastfeeding Self Efficacy of Mothers in Cesarean Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Nursing123
Record Dates: First submitted 2022-12-21; First posted 2023-01-26 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-12

CONDITIONS: Nurse's Role; Breastfeeding
Keywords: skin-to-skin contact; cesarean; newborn; breastfeeding self-efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: intervention group and control group, randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (skin-to-skin contact group) (Experimental): skin-to-skin contact: It is the laying of the newborn in the prone position on the mother's bare chest area with only a diaper on.
  Interventions: Behavioral: Skin-to-Skin contact.
- control group (No Intervention): The routine applications of the hospital were applied to the pregnant women in the control group.

INTERVENTIONS:
Behavioral: Skin-to-Skin contact. — Skin to skin contact: It is the laying of the newborn in the prone position on the mother's bare chest with only a diaper on.
  Arms: intervention group (skin-to-skin contact group)

SUMMARY:
Due to the separation of the mother and the baby after the cesarean section, initiation of breastfeeding by the mother of the newborn in the first hour of life is delayed. The rate of cesarean section in Turkey has increased to 52%, according to the 2019 data of the Center for Disease Control and Prevention, the rate of cesarean section has increased to 31.7% in the world and up to 65% in the USA. It has been reported in the literature that cesarean deliveries are performed with general, spinal and epidural anesthesia types, and the Apgar scores of newborns after cesarean section performed with spinal and epidural anesthesia are high. In this context, the nurse has a key role in initiating and maintaining breastfeeding after early SSC between the mother and the newborn within the first hour following the cesarean section performed with spinal anesthesia. In the literature, there are studies reporting that skin-to-skin contact applied after normal delivery increases the sucking success of newborns, the successful breastfeeding rate, and the rate of exclusive breastfeeding. There are studies examining the effect of early skin-to-skin contact applied after cesarean section on the suckling success of the newborn and only breastfeeding. Breastfeeding self-efficacy refers to a woman's confidence in her ability to breastfeed her baby. It is reported in the literature that skin-to-skin contact and only breastfeeding education have an effect on breastfeeding self-efficacy.

DETAILED DESCRIPTION:
Type of the research: The research was conducted in a randomized controlled experimental type. Mothers and newborns who met the inclusion criteria were randomly selected by tossing a coin and assigned to the intervention or control groups. The data were collected by the researcher by face-to-face interview method.

Independent variable: Skin-to-skin contact. Dependent variables: Sucking efficacy of newborns and breastfeeding self-efficacy of mothers.

Research Hypotheses; H1: Skin-to-skin contact applied after cesarean deliveries performed with spinal anesthesia has an effect on the sucking efficiency of newborns.

H2: Skin-to-skin contact applied after cesarean section with spinal anesthesia has an effect on breastfeeding self-efficacy of mothers

It was performed with a total of 72 women and newborns (37 interventions, 35 control groups) who had a cesarean section with spinal anesthesia in a Training and Research Hospital Gynecology Service in the West of Turkey.

Data were collected using the "Newborn and Parent Information Form", "Breastfeeding Self-Efficacy Short Form Scale" and "LATCH Scale".

ELIGIBILITY:
Inclusion Criteria:

Mothers;

* Planning of cesarean section with spinal anesthesia
* Being between the ages of 18- 45
* Having a singleton pregnancy
* Gestational week is between 37-40 weeks
* Absence of any known health problems (diabetes, gestational diabetes, hypertension, preeclampsia, renal failure, cardiac problems, psychiatric disorders, etc.)
* Agreeing to participate in the study
* Before the skin-to-skin contact procedure, their general condition and vital signs should be checked to be stable
* Being a resident of Kütahya

Newborns (0-28 days);

* Gestational age between 37-40 weeks
* Birth weight between 2500-4500 g
* 1.-5. minute Apgar Score ≥ 7
* Absence of any health problems, anomalies or congenital diseases
* Absence of obstacles to sucking such as frenulum (tongue-tie) or palate problem

Exclusion Criteria:

-

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
The effect of skin-to-skin contact on breastfeeding self efficacy of mothers | through study completion, an average of 1 year
  "Breastfeeding Self-Efficacy Scale Short Form" was used to determine mothers' breastfeeding self-efficacy.
  A high score from the scale indicates that the mother's breastfeeding self-efficacy is high.
The effect of skin-to-skin contact on breastfeeding success of mothers and sucking success of newborns. | through study completion, an average of 1 year
  "LATCH Breastfeeding Diagnostic Scale" was used to determine the effect of skin-to-skin contact on breastfeeding success of mothers and breastfeeding success of newborns. A high score from the scale shows that mothers have good breastfeeding success and newborns have good sucking success.
  The name of the "LATCH Breastfeeding Diagnostic Scale" consists of the English initials of the 5 assessment criteria; [L (Latch on the breast), A (Audible swallowing), T (Type of the nipple), C (Comfort breast/nipple), H (Hold)].

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)